CLINICAL TRIAL: NCT03078556
Title: An Open-label, Randomized, Single Dose, Crossover, Pivotal Bioequivalence Study of Fixed-dose Combination Tablets of Dolutegravir and Lamivudine Versus Dolutegravir and Lamivudine Single Entities and Food Effect Assessment in Healthy Volunteers
Brief Title: Bioequivalence Study of Fixed Dose Versus Single Entities of Dolutegravir and Lamivudine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 204994
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2018-08

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: FDC; Lamivudine; Bio-equivalence; Dolutegravir; HIV
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment sequence A/B: Part 1 (Experimental): Eligible subjects will be randomized in sequence A/B and will receive A: DTG 50 milligram (mg) and 3TC 300 mg single entities in Period 1, B: DTG 3TC FDC formulation 1 tablet in Period 2.
  Interventions: Drug: Dolutegravir; Drug: Lamivudine; Drug: Dolutegravir + Lamivudine FDC Formulation 1
- Treatment sequence B/A: Part 1 (Experimental): Eligible subjects will be randomized in sequence B/A and will receive B: DTG 3TC FDC formulation 1 tablet in Period 1 and A: DTG 50 mg and 3TC 300 mg single entities in Period 2.
  Interventions: Drug: Dolutegravir; Drug: Lamivudine; Drug: Dolutegravir + Lamivudine FDC Formulation 1
- Subjects receiving high fat meal: Part 1 (Experimental): Eligible subjects will be administered single dose of DTG 3TC FDC formulation 1 tablet with high fat meal in Period 3 to study the effect of food on tablet.
  Interventions: Drug: Dolutegravir + Lamivudine FDC Formulation 1
- Treatment sequence A/C: Part 2 (Experimental): Eligible subjects will be randomized in sequence A/B and will receive A: DTG 50 mg and 3TC 300 mg single entities in Period 1 and C: DTG 3TC FDC formulation 2 tablet in Period 2.
  Interventions: Drug: Dolutegravir; Drug: Lamivudine; Drug: Dolutegravir + Lamivudine FDC Formulation 2
- Treatment sequence C/A: Part 2 (Experimental): Eligible subjects will be randomized in sequence C/A and will receive C: DTG 3TC FDC formulation 2 tablet in Period 1 and A: DTG 50 milligram (mg) and 3TC 300 mg single entities in Period 2.
  Interventions: Drug: Dolutegravir; Drug: Lamivudine; Drug: Dolutegravir + Lamivudine FDC Formulation 2
- Subjects receiving high fat meal: Part 2 (Experimental): Eligible subjects will be administered single dose of DTG 3TC FDC formulation 2 tablet with high fat meal in Period 3 to study the effect of food on tablet.
  Interventions: Drug: Dolutegravir + Lamivudine FDC Formulation 2

INTERVENTIONS:
Drug: Dolutegravir — Single dose of DTG 50 mg tablet along with 3TC (EPIVIR) tablet will be given to randomized subjects in parts 1 and 2 with 240 mL of room temperature water. DTG will be a white, film coated, round tablet engraved with SV 572 on one side and 50 on the other side.
  Arms: Treatment sequence A/B: Part 1; Treatment sequence A/C: Part 2; Treatment sequence B/A: Part 1; Treatment sequence C/A: Part 2
Drug: Lamivudine — Single dose 3TC (commercial name: EPIVIR) 300 mg tablet along with DTG tablet will be given to randomized subjects in parts 1 and 2 with 240 mL of room temperature water.<br>3TC will be gray, diamond shaped tablet, engraved "GX EJ7" on one side and plain on the other side.
  Arms: Treatment sequence A/B: Part 1; Treatment sequence A/C: Part 2; Treatment sequence B/A: Part 1; Treatment sequence C/A: Part 2
Drug: Dolutegravir + Lamivudine FDC Formulation 1 — Single dose of DTG 50 mg combined with 3TC 300 mg in a FDC formulation 1 tablet will be administered to randomized subjects in treatment periods 1 and 2 (under fasted state) of Part 1 and the first 16 subjects in treatment period 3 (under fed) of Part 1 with 240 mL of room temperature water. <br>FDC formulation 1 tablets will be oval, biconvex, white, film coated tablet engraved 'SV H7I' on one face.
  Arms: Subjects receiving high fat meal: Part 1; Treatment sequence A/B: Part 1; Treatment sequence B/A: Part 1
Drug: Dolutegravir + Lamivudine FDC Formulation 2 — Single dose of DTG 50 mg combined with 3TC 300 mg in a FDC formulation 2 tablet will be administered to randomized subjects in treatment periods 1 and 2 (under fasted state) and the first 16 subjects in treatment period 3 (under fed) of Part 2 with 240 mL of room temperature water. <br>FDC formulation 2 tablets will be oval, biconvex, white, film coated tablet engraved 'SV 13N' on one face.
  Arms: Subjects receiving high fat meal: Part 2; Treatment sequence A/C: Part 2; Treatment sequence C/A: Part 2

SUMMARY:
This study aims to compare the bioequivalence of two experimental fixed dose combination (FDC) tablets versus single entity products of dolutegravir (DTG) and lamivudine (3TC) in healthy adult subjects. The study will be carried out in two parts. Part 1 of the study will be open label, up to 3 periods design with a wash out period of at least 7 days between treatment periods. Subjects will be randomized to receive either single entities or formulation 1 FDC of DTG and 3TC in a crossover manner in first 2 periods. The first 16 subjects who complete the first two treatment periods and consent to continue will receive a single dose of FDC formulation 1 tablet administered with a high fat meal for a third treatment period. In Part 2 of the study, subjects will be randomized to receive either single entities or formulation 2 FDC of DTG and 3TC in a crossover manner in first 2 periods. Similarly the first 16 subjects will then receive FDC formulation 2 tablets with high fat meal in treatment period 3. Subjects will have a follow-up visit within 7-14 days after the last dose of study drug. Approximately 76 healthy subjects will be included in Part 1 of the study and if Part 2 of the study is conducted, another 76 healthy subjects will be included. The total duration will be approximately 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac evaluation (history, electrocardiogram [ECG]).
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator, in consultation with the Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Subject must be able to swallow 2 tablets at the same time (Reference tablets only).
* Body weight >=50 kilogram (kg) for men and >=45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg per meter square (kg/m^2).
* Male or Female. Female subject: is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: 1. non-reproductive potential defined as: pre-menopausal females with one of the following: documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; hysterectomy; documented bilateral Oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea; in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. 2. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until at least five terminal half-lives OR until any continuing pharmacologic effect has ended, whichever is longer after the last dose of study medication and completion of the follow-up visit.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percentage).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) > 450 milliseconds (msec).
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and ViiV Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces [360 milliliter (mL)] of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 1 month prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Creatinine clearance (CrCL) <90 mL/minute.
* A positive hepatitis B surface antigen (HBsAg) or a positive hepatitis B core antibody with a negative hepatitis B surface antibody, positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood product in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts (Part 1 and Part 2) at a single center in the United States from 27-March-2017 to 18-August-2017 and 154 participants (78 in Part 1 and 76 in Part 2) were randomized. First 16 participants completing the first 2 dosing periods, returned for a 3rd treatment period and received single dose of FDC with high fat meal
Pre-assignment Details: A total of 283 (Part 1: 150, Part 2: 133) participants were screened for this study; 125 (Part 1: 72, Part2: 53) participants were screen failures (SF) and 4 participants were reserved but not used. The reasons for SF: inclusion/exclusion criteria not met (105), withdrew consent (18), physician decision (2).
Groups:
- Part 1:DTG+EPIVIR/DTG+3TC Monolayer/DTG+3TC Monolayer-fed: Participants were randomized to receive dolutegravir (DTG) 50 milligram (mg) tablet plus a single lamivudine (3TC) tablet in Period 1 followed by DTG 50 mg/3TC 300 mg fixed dose combination (FDC) monolayer formulation in Period 2. The first 16 participants who completed treatment periods 1 and 2, received a single dose of the FDC monolayer tablet formulation administered with a high fat meal in Period 3. There was a washout of 7 days between treatment periods.
- Part 1:DTG+3TC Monolayer/DTG+EPIVIR/DTG+3TC Monolayer-fed: Participants were randomized to receive DTG 50 mg/3TC 300 mg FDC monolayer formulation in Period 1 followed by DTG 50 mg tablet plus a single 3TC tablet in Period 2. The first 16 participants who completed treatment periods 1 and 2, received a single dose of the FDC monolayer tablet formulation administered with a high fat meal in Period 3. There was a washout of 7 days between treatment periods.
- Part 2:DTG+EPIVIR/DTG+3TC Bilayer/DTG+3TC Bilayer-fed: Participants were randomized to receive DTG 50 mg tablet plus a single 3TC tablet in Period 1 followed by DTG 50 mg/3TC 300 mg FDC bilayer formulation in Period 2. The first 16 participants who completed treatment periods 1 and 2, received a single dose of the FDC bilayer tablet formulation administered with a high fat meal in Period 3. There was a washout of 7 days between treatment periods.
- Part 2:DTG+3TC Bilayer/DTG+EPIVIR /DTG+3TC Bilayer-fed: Participants were randomized to receive DTG 50 mg/3TC 300 mg FDC bilayer formulation in Period 1 followed by DTG 50 mg tablet plus a single 3TC tablet in Period 2. The first 16 participants who completed treatment periods 1 and 2, received a single dose of the FDC bilayer tablet formulation administered with a high fat meal in Period 3. There was a washout of 7 days between treatment periods.
Period: Treatment Period 1 (4 Days)
Arm/Group | Part 1:DTG+EPIVIR/DTG+3TC Monolayer/DTG+3TC Monolayer-fed | Part 1:DTG+3TC Monolayer/DTG+EPIVIR/DTG+3TC Monolayer-fed | Part 2:DTG+EPIVIR/DTG+3TC Bilayer/DTG+3TC Bilayer-fed | Part 2:DTG+3TC Bilayer/DTG+EPIVIR /DTG+3TC Bilayer-fed
Started | 39 | 39 | 38 | 38
Completed | 39 | 38 | 38 | 38
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | Part 1:DTG+EPIVIR/DTG+3TC Monolayer/DTG+3TC Monolayer-fed | Part 1:DTG+3TC Monolayer/DTG+EPIVIR/DTG+3TC Monolayer-fed | Part 2:DTG+EPIVIR/DTG+3TC Bilayer/DTG+3TC Bilayer-fed | Part 2:DTG+3TC Bilayer/DTG+EPIVIR /DTG+3TC Bilayer-fed
Started | 39 | 38 | 38 | 38
Completed | 37 | 36 | 37 | 37
Not Completed | 2 | 2 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Period: Treatment Period 2 (4 Days)
Arm/Group | Part 1:DTG+EPIVIR/DTG+3TC Monolayer/DTG+3TC Monolayer-fed | Part 1:DTG+3TC Monolayer/DTG+EPIVIR/DTG+3TC Monolayer-fed | Part 2:DTG+EPIVIR/DTG+3TC Bilayer/DTG+3TC Bilayer-fed | Part 2:DTG+3TC Bilayer/DTG+EPIVIR /DTG+3TC Bilayer-fed
Started | 37 | 36 | 37 | 37
Completed | 37 | 36 | 37 | 37
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | Part 1:DTG+EPIVIR/DTG+3TC Monolayer/DTG+3TC Monolayer-fed | Part 1:DTG+3TC Monolayer/DTG+EPIVIR/DTG+3TC Monolayer-fed | Part 2:DTG+EPIVIR/DTG+3TC Bilayer/DTG+3TC Bilayer-fed | Part 2:DTG+3TC Bilayer/DTG+EPIVIR /DTG+3TC Bilayer-fed
Started | 9 | 7 | 7 | 9
Completed | 9 | 7 | 7 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3 (4 Days)
Arm/Group | Part 1:DTG+EPIVIR/DTG+3TC Monolayer/DTG+3TC Monolayer-fed | Part 1:DTG+3TC Monolayer/DTG+EPIVIR/DTG+3TC Monolayer-fed | Part 2:DTG+EPIVIR/DTG+3TC Bilayer/DTG+3TC Bilayer-fed | Part 2:DTG+3TC Bilayer/DTG+EPIVIR /DTG+3TC Bilayer-fed
Started | 9 | 7 | 7 | 9
Completed | 9 | 7 | 7 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who enrolled in the study and received at least one dose of study drug.
Groups:
- Part 1: Participants were randomized into treatment sequence A/B (treatment A in Period 1 followed by B in Period 2) or B/A (treatment B in Period 1 followed by A in Period 2), where A=dolutegravir (DTG) 50 milligram (mg) tablet plus a single lamivudine (3TC) tablet and treatment B= DTG 50 mg/3TC 300 mg fixed dose combination (FDC) monolayer formulation. The first 16 participants who completed treatment periods 1 and 2, received a single dose of the FDC monolayer tablet formulation administered with a high fat meal in Period 3. There was a washout period of at least 7 days between each treatment period. In treatment periods 1 and 2, single dose of the treatments were administered in the fasted state.
- Part 2: Participants were randomized into treatment sequence A/C (treatment A in Period 1 followed by C in Period 2) or C/A (treatment C in Period 1 followed by A in Period 2), where A=DTG 50 mg tablet plus a single 3TC tablet and treatment C= DTG 50 mg/3TC 300 mg FDC bilayer formulation. The first 16 participants who completed treatment periods 1 and 2, received a single dose of the FDC bilayer tablet formulation administered with a high fat meal in Period 3. There was a washout period of at least 7 days between each treatment period.
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 78 | 76 | 154
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.4 (9.37) | 31.6 (11.18) | 30.5 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 53 | 50 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 1 | 7
  Asian- Central/South Asian Heritage | 1 | 1 | 2
  Asian- East Asian Heritage | 0 | 1 | 1
  Asian- South East Asian Heritage | 1 | 0 | 1
  Black or African American | 20 | 23 | 43
  White-White/Caucasian/European Heritage | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity [AUC (0-Inf)] of Plasma DTG and 3TC in the Fasted State: Part 1
Description: Blood samples were collected at indicated time points to study the pharmacokinetic (PK) profile of DTG and 3TC when administered as FDC tablet compared to co-administration of separate tablet formulations of DTG and 3TC in fasted state. The 4-hour post-dose sample was drawn prior to the participant's first post-dose meal. At each time point, 2 mL of blood was collected. PK parameters of monolayer FDC tablet formulation of DTG and 3TC was evaluated under fasted condition in Periods 1 and 2 of Part 1.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter Bioequivalence (BE) Summary Population comprised of all participants who have evaluable PK parameters for both analytes and for both Period 1 and Period 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Groups:
- A: DTG 50 mg + EPIVIR 300 mg: Participants received a single oral dose of DTG 50 mg and EPIVIR 300 mg tablet(s) at the same time with 240 mL of water in Periods 1 and 2 of Part 1. Treatments were administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
- B: DTG 50 mg/ 3TC 300 mg Monolayer FDC: Participants received a single oral dose of DTG 50 mg and 3TC 300 mg monolayer FDC tablet formulation in Periods 1 and 2 of Part 1. Treatment was administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Hour*micrograms per milliliter
  DTG | 43.1456 (39.29) | 54.8793 (31.60)
  3TC | 12.3337 (19.88) | 12.7603 (19.77)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 1.2710, 90% CI 2-sided [1.1894 to 1.3582] — Ratio (B/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 1.0341, 90% CI 2-sided [1.0097 to 1.0591] — Ratio (B/A) of plasma 3TC has been presented

2. Primary Outcome: AUC (0-Inf) of Plasma DTG and 3TC in the Fasted State: Part 2
Description: Blood samples were collected at given time points to study the PK profile of DTG and 3TC when administered as FDC tablet compared to co-administration of separate tablet formulations of DTG and 3TC in fasted state. The 4-hour post-dose sample was drawn prior to the participant's first post-dose meal. At each time point, 2 mL of blood was collected. PK parameters of bilayer FDC tablet formulation of DTG and 3TC was evaluated under fasted conditions in Periods 1 and 2 of Part 2.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population. Only those participants with data available at the specified data points were analyzed, represented by n= X,X in the category titles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- A: DTG 50 mg + EPIVIR 300 mg: Participants received a single oral dose of DTG 50 mg and EPIVIR 300 mg tablet(s) at the same time with 240 mL of water in Periods 1 and 2 of Part 2. Treatments were administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
- C: DTG 50 mg/ 3TC 300 mg Bilayer FDC: Participants received a single oral dose of DTG 50 mg and 3TC 300 mg bilayer FDC tablet formulation in Periods 1 and 2 of Part 2. Treatment was administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Hours*micrograms per milliliter
  DTG, n= 74,74 | 47.2391 (40.29) | 54.5594 (32.12)
  3TC, n= 73,74: number analyzed (Participants) | 73 | 74
  3TC, n= 73,74 | 12.7713 (18.63) | 13.5624 (17.94)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 1.1550, 90% CI 2-sided [1.0699 to 1.2468] — Ratio (C/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 1.0635, 90% CI 2-sided [1.0413 to 1.0861] — Ratio (C/A) of plasma 3TC has been presented

3. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to the Last Quantifiable Time Point (AUC[0-t]) of Plasma DTG and 3TC in the Fasted State: Part 1
Description: Blood samples were collected at indicated time points to study the PK profile of DTG and 3TC when administered as FDC tablet compared to co-administration of separate tablet formulations of DTG and 3TC in fasted state. The 4-hour post-dose sample was drawn prior to the participant's first post-dose meal. At each time point, 2 mL of blood was collected. PK parameters of monolayer FDC tablet formulation of DTG and 3TC was evaluated under fasted condition in Periods 1 and 2 of Part 1.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Hours*micrograms per milliliter
  DTG | 41.4207 (39.36) | 52.8754 (31.16)
  3TC | 12.1571 (20.19) | 12.6147 (19.75)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 1.2756, 90% CI 2-sided [1.1919 to 1.3651] — Ratio (B/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 1.0372, 90% CI 2-sided [1.0116 to 1.0634] — Ratio (B/A) of plasma 3TC has been presented

4. Primary Outcome: AUC(0-t) of Plasma DTG and 3TC in the Fasted State: Part 2
Description: Blood samples were collected at indicated time points to study the PK profile of DTG and 3TC when administered as FDC tablet compared to co-administration of separate tablet formulations of DTG and 3TC in fasted state. The 4-hour post-dose sample was drawn prior to the participant's first post-dose meal. At each time point, 2 mL of blood was collected. PK parameters of bilayer FDC tablet formulation of DTG and 3TC was evaluated under fasted condition in Periods 1 and 2 of Part 2.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram/milliliter
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Hour*microgram/milliliter
  DTG | 45.2043 (39.57) | 52.3372 (31.46)
  3TC | 12.4790 (19.19) | 13.3552 (18.10)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 1.1578, 90% CI 2-sided [1.0718 to 1.2507] — Ratio (C/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 1.0702, 90% CI 2-sided [1.0464 to 1.0946] — Ratio (C/A) of plasma 3TC has been presented

5. Primary Outcome: Maximum Observed Concentration (Cmax) of Plasma DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Groups:
- B: DTG 50 mg/ 3TC 300 mg Monolayer FDC: Participants received a single oral dose of DTG 50 mg and 3TC 300 mg monolayer FDC tablet formulation in Periods 1 and 2 of Part 1. Treatments were administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Micrograms per milliliter
  DTG | 2.4065 (38.95) | 3.0817 (31.86)
  3TC | 2.6650 (29.04) | 3.1885 (28.07)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 1.2805, 90% CI 2-sided [1.1890 to 1.3790] — Ratio (B/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 1.1956, 90% CI 2-sided [1.1437 to 1.2498] — Ratio (B/A) of plasma 3TC has been presented

6. Primary Outcome: Cmax of Plasma DTG and 3TC in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Groups:
- B: DTG 50 mg/ 3TC 300 mg Bilayer FDC: Participants received a single oral dose of DTG 50mg and 3TC 300mg bilayer FDC tablet formulation in Periods 1 and 2 of Part 2. Treatment was administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Micrograms per milliliter
  DTG | 2.5531 (36.38) | 2.9132 (30.55)
  3TC | 2.4428 (28.25) | 3.2185 (29.30)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 1.1410, 90% CI 2-sided [1.0533 to 1.2361] — Ratio (C/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 1.3176, 90% CI 2-sided [1.2616 to 1.3760] — Ratio (C/A) of plasma 3TC has been presented

7. Secondary Outcome: Absorption Lag Time (Tlag) of DTG and 3TC in Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Hour
  DTG | 0.0000 [0.0000 to 0.756] | 0.0000 [0.0000 to 0.261]
  3TC | 0.0000 [0.0000 to 0.252] | 0.0000 [0.0000 to 0.261]
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [0.000 to 0.000] — Median Difference of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [0.000 to 0.000] — Median Difference of plasma 3TC has been presented

8. Secondary Outcome: Tlag of DTG and 3TC in Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Hour
  DTG | 0.0000 [0.0000 to 0.261] | 0.0000 [0.0000 to 0.266]
  3TC | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.252]
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [-0.004 to 0.000] — Median Difference of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [0.000 to 0.000] — Median Difference of plasma 3TC has been presented

9. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Hour
  DTG | 2.0072 [0.500 to 8.009] | 2.0017 [0.500 to 5.012]
  3TC | 1.0047 [0.500 to 4.005] | 1.0008 [0.500 to 3.500]
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Median Difference (Final Values) = -0.127, 90% CI 2-sided [-0.500 to 0.248] — Median Difference of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Median Difference (Final Values) = -0.126, 90% CI 2-sided [-0.253 to -0.001] — Median Difference of plasma 3TC has been presented

10. Secondary Outcome: Tmax of DTG and 3TC in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Hour
  DTG | 2.5008 [0.500 to 5.011] | 2.5004 [0.500 to 6.001]
  3TC | 1.0063 [0.500 to 4.002] | 1.0011 [0.500 to 3.501]
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Median Difference (Final Values) = -0.127, 90% CI 2-sided [-0.497 to 0.132] — Median Difference of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Median Difference (Final Values) = -0.248, 90% CI 2-sided [-0.376 to -0.001] — Median Difference of plasma 3TC has been presented

11. Secondary Outcome: Time of the Last Quantifiable Concentration (Tlast) of DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Hour
  DTG | 72.0031 [48.000 to 74.636] | 71.9303 [48.003 to 76.236]
  3TC | 71.9289 [47.673 to 74.636] | 71.9303 [70.790 to 76.236]

12. Secondary Outcome: Tlast of DTG and 3TC in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Hour
  DTG | 71.6813 [48.006 to 75.301] | 71.8243 [71.005 to 72.632]
  3TC | 71.7138 [48.000 to 75.301] | 71.8153 [48.007 to 72.632]

13. Secondary Outcome: Time to Reach Half the Maximum Plasma Concentration (t1/2) of DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Hour
  DTG | 14.6917 [10.575 to 21.375] | 14.7557 [10.461 to 21.392]
  3TC | 17.0395 [8.281 to 34.542] | 17.3436 [12.436 to 34.675]

14. Secondary Outcome: t1/2 of DTG and 3TC in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population. Only those participants with data available at the specified time points were analyzed indicated by n=X in category titles.
Measure: Median (Full Range); unit: Hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Hour
  DTG, n= 74,74 | 15.1538 [9.711 to 21.966] | 14.7893 [9.815 to 21.486]
  3TC, n= 73,74: number analyzed (Participants) | 73 | 74
  3TC, n= 73,74 | 17.8421 [10.195 to 47.171] | 18.1071 [7.367 to 48.613]

15. Secondary Outcome: Apparent Elimination Rate Constant (Lambda z) of DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Median (Full Range); unit: Per hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Per hour
  DTG | 0.0472 [0.032 to 0.066] | 0.0470 [0.032 to 0.066]
  3TC | 0.0407 [0.020 to 0.084] | 0.0400 [0.020 to 0.056]

16. Secondary Outcome: Lambda z of DTG and 3TC in in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population. Only those participants with data available at the specified data points were analyzed (represented by n= X,X in the category titles).
Measure: Median (Full Range); unit: Per hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Per hour
  DTG, n=74,74 | 0.0457 [0.032 to 0.071] | 0.0469 [0.032 to 0.071]
  3TC, n= 73,74: number analyzed (Participants) | 73 | 74
  3TC, n= 73,74 | 0.0388 [0.015 to 0.068] | 0.0383 [0.014 to 0.094]

17. Secondary Outcome: Percentage of Extrapolated AUC (0 to Inf) of DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population.
Measure: Median (Full Range); unit: Percentage of AUC
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Percentage of AUC
  DTG | 3.4967 [1.015 to 15.084] | 3.2582 [0.908 to 9.967]
  3TC | 1.0287 [0.343 to 7.305] | 0.9052 [0.428 to 5.334]

18. Secondary Outcome: Percentage of Extrapolated AUC(0 to Inf) of DTG and 3TC in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 14
Measure: Median (Full Range); unit: Percentage of AUC
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Percentage of AUC
  DTG, n= 74,74 | 3.8923 [0.932 to 10.512] | 3.5773 [0.659 to 9.570]
  3TC, n= 73,74: number analyzed (Participants) | 73 | 74
  3TC, n= 73,74 | 1.2518 [0.344 to 6.409] | 1.1432 [0.394 to 7.867]

19. Secondary Outcome: AUC of 0 to 24 Hours (AUC[0-24]) of DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Hours*microgram per milliliter
  DTG | 29.4257 (38.40) | 37.6112 (30.28)
  3TC | 11.3960 (20.92) | 11.9418 (20.09)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 1.2774, 90% CI 2-sided [1.1931 to 1.3676] — Ratio (B/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 1.0475, 90% CI 2-sided [1.0185 to 1.0773] — Ratio (B/A) of plasma 3TC has been presented

20. Secondary Outcome: AUC(0-24) of DTG and 3TC in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Hours*microgram per milliliter
  DTG | 31.5664 (37.73) | 36.6126 (30.93)
  3TC | 11.6419 (20.23) | 12.5810 (18.50)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 1.1599, 90% CI 2-sided [1.0711 to 1.2560] — Ratio (C/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 1.0807, 90% CI 2-sided [1.0539 to 1.1081] — Ratio (C/A) of plasma 3TC has been presented

21. Secondary Outcome: Apparent Oral Clearance (CL/F) of DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Liters per hour
  DTG | 1.1589 (39.29) | 0.9111 (31.60)
  3TC | 24.3236 (19.88) | 23.5104 (19.77)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 0.7868, 90% CI 2-sided [0.7363 to 0.8408] — Ratio (B/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 0.9670, 90% CI 2-sided [0.9442 to 0.9904] — Ratio (B/A) of plasma 3TC has been presented

22. Secondary Outcome: CL/F of DTG and 3TC in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population. Only those participants with data available at the specified time points were analyzed represented by n=X in the category titles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Liters per hour
  DTG, n= 74, 74 | 1.0584 (40.29) | 0.9164 (32.12)
  3TC, n= 73, 74: number analyzed (Participants) | 73 | 74
  3TC, n= 73, 74 | 23.4901 (18.63) | 22.1200 (17.94)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 0.8658, 90% CI 2-sided [0.8021 to 0.9347] — Ratio (C/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 0.9403, 90% CI 2-sided [0.9207 to 0.9604] — Ratio (C/A) of plasma 3TC has been presented

23. Secondary Outcome: Apparent Oral Volume of Distribution (Vz/F) of DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Liters
  DTG | 24.6254 (37.80) | 19.3399 (30.05)
  3TC | 616.7365 (34.52) | 598.8651 (29.07)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 0.7859, 90% CI 2-sided [0.7318 to 0.8440] — Ratio (B/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 0.9704, 90% CI 2-sided [0.9157 to 1.0284] — Ratio (B/A) of plasma 3TC has been presented

24. Secondary Outcome: Vz/F of DTG and 3TC in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Liters
  DTG, n= 74, 74 | 23.1159 (37.18) | 19.8124 (32.73)
  3TC, n= 73, 74: number analyzed (Participants) | 73 | 74
  3TC, n= 73, 74 | 650.7952 (35.55) | 599.5525 (34.28)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 0.8571, 90% CI 2-sided [0.7914 to 0.9282] — Ratio (C/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 0.9153, 90% CI 2-sided [0.8613 to 0.9728] — Ratio (C/A) of plasma 3TC has been presented

25. Secondary Outcome: Concentration at 24 Hours Post-dose (C24) of DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Micrograms per milliliter
  DTG | 0.6373 (40.18) | 0.8059 (32.77)
  3TC | 0.0331 (32.13) | 0.0318 (31.81)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 1.2632, 90% CI 2-sided [1.1811 to 1.3511] — Ratio (B/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 0.9598, 90% CI 2-sided [0.9268 to 0.9941] — Ratio (B/A) of plasma 3TC has been presented

26. Secondary Outcome: C24 of DTG and 3TC in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Micrograms per milliliter
  DTG | 0.7065 (41.48) | 0.8071 (33.83)
  3TC | 0.0366 (30.39) | 0.0350 (31.19)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 1.1425, 90% CI 2-sided [1.0597 to 1.2317] — Ratio (C/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 0.9548, 90% CI 2-sided [0.9299 to 0.9804] — Ratio (C/A) of plasma 3TC has been presented

27. Secondary Outcome: Last Quantifiable Concentration (Clast) of DTG and 3TC in the Fasted State: Part 1
Description: as for outcome 3
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC
Number analyzed (Participants) | 73 | 73
Micrograms per milliliter
  DTG | 0.0702 (58.85) | 0.0832 (56.42)
  3TC | 0.0056 (43.03) | 0.0050 (37.58)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 1.1839, 90% CI 2-sided [1.0921 to 1.2834] — Ratio (B/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs B: DTG 50 mg/ 3TC 300 mg Monolayer FDC; Test type: Other; Ratio = 0.8874, 90% CI 2-sided [0.8340 to 0.9443] — Ratio (B/A) of plasma 3TC has been presented

28. Secondary Outcome: Clast of DTG and 3TC in the Fasted State: Part 2
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter BE Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | A: DTG 50 mg + EPIVIR 300 mg | C: DTG 50 mg/ 3TC 300 mg Bilayer FDC
Number analyzed (Participants) | 74 | 74
Micrograms per milliliter
  DTG | 0.0800 (66.94) | 0.0862 (65.26)
  3TC | 0.0069 (47.83) | 0.0062 (41.60)
Statistical Analysis 1: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 1.0780, 90% CI 2-sided [0.9958 to 1.1670] — Ratio (B/A) of plasma DTG has been presented
Statistical Analysis 2: Comparison: A: DTG 50 mg + EPIVIR 300 mg vs C: DTG 50 mg/ 3TC 300 mg Bilayer FDC; Test type: Other; Ratio = 0.9049, 90% CI 2-sided [0.8474 to 0.9663] — Ratio (B/A) of plasma 3TC has been presented

29. Secondary Outcome: AUC (0-Inf) of Plasma DTG and 3TC in the Fed State: Part 1
Description: Blood samples for PK analysis of DTG and 3TC were collected at given time points to study the PK profile of DTG and 3TC FDC tablet(s). The 4-hour post-dose sample was drawn prior to the participant's first post-dose meal. At each time point, 2 mL of blood was collected. The effect of food on DTG and 3TC monolayer FDC tablet formulations was assessed in Period 3 of Part 1.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter food effect (FD) Summary Population comprised of participants who participated in the food effect part of the study and had evaluable PK parameters for both fed and fasted administration of the FDC tablet formulation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Bfed: DTG 50 mg/3TC 300 mg Monolayer FDC Fed: Participants received DTG 50 mg and 3TC 300 mg monolayer FDC tablet formulation (Product Code AH). Treatment was administered with high fat meal. There was a washout period of at least 7 days (-4 hours) between each dose of the study drug.
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg/3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hours*microgram per milliliter
  DTG | 62.3435 (32.34) | 71.9777 (19.99)
  3TC | 13.4357 (21.02) | 12.8668 (18.50)
Statistical Analysis 1: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg/3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 1.1545, 90% CI 2-sided [1.0208 to 1.3058] — Ratio (Bfed/B) of plasma DTG has been presented
Statistical Analysis 2: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg/3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 0.9577, 90% CI 2-sided [0.9126 to 1.0049] — Ratio (Bfed/B) of plasma 3TC has been presented

30. Secondary Outcome: AUC (0-Inf) of Plasma DTG and 3TC in the Fed State: Part 2
Description: Blood samples for PK analysis of DTG and 3TC were collected at given time points to study the PK profile of DTG and 3TC FDC tablet(s). The 4-hour post-dose sample was drawn prior to the participant's first post-dose meal. At each time point, 2 mL of blood was collected. The effect of food on DTG and 3TC bilayer FDC tablet formulations was assessed in Period 3 of Part 2.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- C: DTG 50 mg and 3TC 300 mg Bilayer FDC: Participants received a single oral dose of DTG 50 mg and 3TC 300 mg bilayer FDC tablet formulation in Periods 1 and 2 of Part 2. Treatment was administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
- Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed: Participants received a single oral dose of DTG 50 mg and 3TC 300 mg bilayer FDC tablet formulation along with a high fat meal in Period 3 of Part 2.
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hours*microgram per milliliter
  DTG | 57.6561 (35.93) | 76.4283 (22.36)
  3TC | 14.6420 (18.50) | 13.3443 (20.34)
Statistical Analysis 1: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 1.3256, 90% CI 2-sided [1.1837 to 1.4845] — Ratio (Cfed/C) of plasma DTG has been presented
Statistical Analysis 2: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 0.9114, 90% CI 2-sided [0.8658 to 0.9593] — Ratio (Cfed/C) of plasma 3TC has been presented

31. Secondary Outcome: AUC (0-t) of Plasma DTG and 3TC in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter
Groups:
- Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed: Participants received DTG 50 mg and 3TC 300 mg monolayer FDC tablet formulation (Product Code AH). Treatment was administered with high fat meal. There was a washout period of at least 7 days (-4 hours) between each dose of the study drug.
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hour*microgram per milliliter
  DTG | 60.3212 (31.78) | 69.2560 (18.92)
  3TC | 13.2818 (20.90) | 12.6491 (18.63)
Statistical Analysis 1: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 1.1481, 90% CI 2-sided [1.0154 to 1.2982] — Ratio (Bfed/B) of plasma DTG has been presented
Statistical Analysis 2: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 0.9524, 90% CI 2-sided [0.9086 to 0.9983] — Ratio (Bfed/B) of plasma 3TC has been presented

32. Secondary Outcome: AUC (0-t) of Plasma DTG and 3TC in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hour*microgram per milliliter
  DTG | 55.2176 (35.33) | 72.7545 (20.22)
  3TC | 14.4706 (18.72) | 13.0923 (20.57)
Statistical Analysis 1: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 1.3176, 90% CI 2-sided [1.1750 to 1.4775] — Ratio (Cfed/C) of plasma DTG has been presented
Statistical Analysis 2: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 0.9048, 90% CI 2-sided [0.8592 to 0.9528] — Ratio (Cfed/C) of plasma 3TC has been presented

33. Secondary Outcome: Cmax of Plasma DTG and 3TC in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Micrograms per milliliter
  DTG | 3.5068 (30.27) | 3.7900 (20.97)
  3TC | 3.5413 (27.14) | 2.5132 (18.74)
Statistical Analysis 1: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 1.0808, 90% CI 2-sided [0.9527 to 1.2261] — Ratio (Bfed/B) of plasma DTG has been presented
Statistical Analysis 2: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 0.7097, 90% CI 2-sided [0.6474 to 0.7779] — Ratio (Bfed/B) of plasma 3TC has been presented

34. Secondary Outcome: Cmax of Plasma DTG and 3TC in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Micrograms per milliliter
  DTG | 3.1015 (35.62) | 3.7516 (21.31)
  3TC | 3.5824 (35.18) | 2.4453 (33.88)
Statistical Analysis 1: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 1.2096, 90% CI 2-sided [1.0521 to 1.3908] — Ratio (Cfed/C) of plasma DTG has been presented
Statistical Analysis 2: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 0.6826, 90% CI 2-sided [0.5861 to 0.7950] — Ratio (Cfed/C) of plasma 3TC has been presented

35. Secondary Outcome: Tlag of DTG and 3TC in Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hour
  DTG | 0.0000 [0.0000 to 0.251] | 0.2522 [0.0000 to 1.000]
  3TC | 0.0000 [0.0000 to 0.251] | 0.0000 [0.0000 to 0.255]
Statistical Analysis 1: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Median Difference (Final Values) = 0.254, 90% CI 2-sided [0.250 to 0.378] — Median Difference of plasma DTG has been presented
Statistical Analysis 2: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Median Difference (Final Values) = 0.125, 90% CI 2-sided [0.000 to 0.127] — Median Difference of plasma 3TC has been presented

36. Secondary Outcome: Tlag of DTG and 3TC in Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hour
  DTG | 0.0000 [0.0000 to 0.258] | 0.1253 [0.0000 to 0.751]
  3TC | 0.0000 [0.0000 to 0.252] | 0.0000 [0.0000 to 0.257]
Statistical Analysis 1: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Median Difference (Final Values) = 0.126, 90% CI 2-sided [0.000 to 0.250] — Median Difference of plasma DTG has been presented
Statistical Analysis 2: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Median Difference (Final Values) = 0.000, 90% CI 2-sided [0.000 to 0.125] — Median Difference of plasma 3TC has been presented

37. Secondary Outcome: Tmax of DTG and 3TC in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hour
  DTG | 1.5013 [0.503 to 5.002] | 5.0006 [2.001 to 12.009]
  3TC | 1.0001 [0.500 to 2.001] | 3.5003 [1.011 to 5.006]
Statistical Analysis 1: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Median Difference (Final Values) = 3.017, 90% CI 2-sided [1.872 to 4.496] — Median Difference of plasma DTG has been presented
Statistical Analysis 2: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Median Difference (Final Values) = 2.113, 90% CI 2-sided [1.500 to 2.751] — Median Difference of plasma 3TC has been presented

38. Secondary Outcome: Tmax of DTG and 3TC in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hour
  DTG | 1.5007 [0.751 to 3.001] | 5.0019 [1.011 to 8.004]
  3TC | 1.0003 [0.503 to 2.506] | 2.7508 [1.001 to 6.001]
Statistical Analysis 1: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Median Difference (Final Values) = 2.500, 90% CI 2-sided [1.748 to 3.751] — Median Difference of plasma DTG has been presented
Statistical Analysis 2: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Median Difference (Final Values) = 1.503, 90% CI 2-sided [0.998 to 2.252] — Median Difference of plasma 3TC has been presented

39. Secondary Outcome: T1/2 of DTG and 3TC in the Fed State: Part 1
Description: Blood samples for PK analysis of DTG and 3TC were collected at given time points to study the PK profile of DTG and 3TC FDC tablet(s). The 4-hour post-dose sample was drawn prior to the participant's first post-dose meal. At each time point, 2 mL of blood. The effect of food on DTG and 3TC monolayer FDC tablet formulations was assessed in Period 3 of Part 1.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hour
  DTG | 14.5843 [12.077 to 16.806] | 14.5816 [10.889 to 17.259]
  3TC | 18.3614 [12.509 to 30.759] | 19.8579 [9.977 to 34.144]

40. Secondary Outcome: T1/2 of DTG and 3TC in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Hour
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hour
  DTG | 14.9828 [11.355 to 20.563] | 15.1718 [12.193 to 19.945]
  3TC | 17.2250 [13.259 to 37.099] | 19.7311 [13.384 to 27.781]

41. Secondary Outcome: Lambda z of DTG and 3TC in in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Per hour
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Per hour
  DTG | 0.0475 [0.041 to 0.057] | 0.0475 [0.040 to 0.064]
  3TC | 0.0378 [0.023 to 0.055] | 0.0349 [0.020 to 0.069]

42. Secondary Outcome: Lambda z of DTG and 3TC in in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Per hour
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Per hour
  DTG | 0.0463 [0.034 to 0.061] | 0.0457 [0.035 to 0.057]
  3TC | 0.0403 [0.019 to 0.052] | 0.0351 [0.025 to 0.052]

43. Secondary Outcome: Clast of DTG and 3TC in in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Micrograms per milliliter
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Micrograms per milliliter
  DTG | 0.1060 [0.035 to 0.180] | 0.1190 [0.043 to 0.243]
  3TC | 0.0048 [0.003 to 0.014] | 0.0066 [0.004 to 0.016]

44. Secondary Outcome: Clast of DTG and 3TC in in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Micrograms per milliliter
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Micrograms per milliliter
  DTG | 0.0975 [0.031 to 0.240] | 0.1310 [0.051 to 0.363]
  3TC | 0.0059 [0.003 to 0.011] | 0.0091 [0.003 to 0.015]

45. Secondary Outcome: Percentage of Extrapolated AUC (0-inf) in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Percentage of AUC
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Percentage of AUC
  DTG | 3.3305 [1.490 to 4.845] | 3.8870 [1.094 to 6.134]
  3TC | 0.8856 [0.561 to 3.510] | 1.4830 [0.788 to 4.324]

46. Secondary Outcome: Percentage of Extrapolated AUC (0-inf) in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Percentage of AUC
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Percentage of AUC
  DTG | 3.6835 [1.069 to 8.601] | 3.8790 [1.561 to 9.126]
  3TC | 1.0443 [0.467 to 3.859] | 1.7467 [0.567 to 3.642]

47. Secondary Outcome: AUC(0-24) of DTG and 3TC in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hour*microgram per milliliter
  DTG | 43.1879 (29.88) | 46.8555 (16.95)
  3TC | 12.6113 (21.25) | 11.8076 (18.71)
Statistical Analysis 1: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 1.0849, 90% CI 2-sided [0.9613 to 1.2245] — Ratio (Bfed/B) of plasma DTG has been presented
Statistical Analysis 2: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 0.9363, 90% CI 2-sided [0.8913 to 0.9836] — Ratio (Bfed/B) of plasma 3TC has been presented

48. Secondary Outcome: AUC(0-24) of DTG and 3TC in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hour*microgram per milliliter
  DTG | 38.6325 (34.53) | 48.2012 (15.53)
  3TC | 13.7012 (19.24) | 12.1065 (21.09)
Statistical Analysis 1: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Median Difference (Final Values) = 1.2477, 90% CI 2-sided [1.1013 to 1.4136] — Median Difference of plasma DTG has been presented
Statistical Analysis 2: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Median Difference (Final Values) = 0.8836, 90% CI 2-sided [0.8351 to 0.9350] — Median Difference of plasma 3TC has been presented

49. Secondary Outcome: CL/F of DTG and 3TC in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Liters per hour
  DTG | 0.8020 (32.34) | 0.6947 (19.99)
  3TC | 22.3285 (21.02) | 23.3159 (18.50)
Statistical Analysis 1: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 0.8661, 90% CI 2-sided [0.7658 to 0.9796] — Ratio (Bfed/B) of plasma DTG has been presented
Statistical Analysis 2: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 1.0442, 90% CI 2-sided [0.9951 to 1.0957] — Ratio (Bfed/B) of plasma 3TC has been presented

50. Secondary Outcome: CL/F of DTG and 3TC in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Liters per hour
  DTG | 0.8672 (35.93) | 0.6542 (22.36)
  3TC | 20.4890 (18.50) | 22.4815 (20.34)
Statistical Analysis 1: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 0.7544, 90% CI 2-sided [0.6736 to 0.8448] — Ratio (Cfed/C) of plasma DTG has been presented
Statistical Analysis 2: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 1.0972, 90% CI 2-sided [1.0424 to 1.1550] — Ratio (Cfed/C) of plasma 3TC has been presented

51. Secondary Outcome: Tlast of DTG and 3TC in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Hours
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hours
  DTG | 71.8265 [71.124 to 72.301] | 71.9758 [71.330 to 72.869]
  3TC | 71.8265 [71.124 to 72.301] | 71.9758 [71.330 to 72.869]

52. Secondary Outcome: Tlast of DTG and 3TC in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Median (Full Range); unit: Hours
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Hours
  DTG | 72.0292 [71.446 to 72.269] | 71.8711 [71.080 to 72.381]
  3TC | 72.0292 [71.446 to 72.269] | 71.8711 [71.080 to 72.381]

53. Secondary Outcome: Vz/F of DTG and 3TC in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Liters
  DTG | 16.7520 (28.45) | 14.4964 (15.87)
  3TC | 593.2054 (29.23) | 643.0977 (41.08)
Statistical Analysis 1: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 0.8654, 90% CI 2-sided [0.7629 to 0.9816] — Ratio (Bfed/B) of plasma DTG has been presented
Statistical Analysis 2: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 1.0841, 90% CI 2-sided [0.9139 to 1.2860] — Ratio (Bfed/B) of plasma 3TC has been presented

54. Secondary Outcome: Vz/F of DTG and 3TC in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Liters
  DTG | 19.0954 (36.45) | 14.6215 (11.63)
  3TC | 535.8125 (35.63) | 641.3744 (32.10)
Statistical Analysis 1: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 0.7657, 90% CI 2-sided [0.6702 to 0.8749] — Ratio (Cfed/C) of plasma DTG has been presented
Statistical Analysis 2: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 1.1970, 90% CI 2-sided [1.0869 to 1.3182] — Ratio (Cfed/C) of plasma 3TC has been presented

55. Secondary Outcome: C24 of DTG and 3TC in the Fed State: Part 1
Description: as for outcome 29
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed
Number analyzed (Participants) | 16 | 16
Micrograms per milliliter
  DTG | 0.9216 (36.08) | 1.1916 (25.03)
  3TC | 0.0304 (33.07) | 0.0366 (35.90)
Statistical Analysis 1: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 1.2929, 90% CI 2-sided [1.1281 to 1.4819] — Ratio (Bfed/B) of plasma DTG has been presented
Statistical Analysis 2: Comparison: B: DTG 50 mg/ 3TC 300 mg Monolayer FDC vs Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed; Test type: Other; Ratio = 1.2015, 90% CI 2-sided [1.1074 to 1.3036] — Ratio (Bfed/B) of plasma 3TC has been presented

56. Secondary Outcome: C24 of DTG and 3TC in the Fed State: Part 2
Description: as for outcome 30
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Parameter FD Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 16 | 16
Micrograms per milliliter
  DTG | 0.8355 (38.46) | 1.2273 (25.73)
  3TC | 0.0350 (39.91) | 0.0417 (38.62)
Statistical Analysis 1: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 1.4690, 90% CI 2-sided [1.3009 to 1.6588] — Ratio (Cfed/C) of plasma DTG has been presented
Statistical Analysis 2: Comparison: C: DTG 50 mg and 3TC 300 mg Bilayer FDC vs Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed; Test type: Other; Ratio = 1.1935, 90% CI 2-sided [1.1142 to 1.2785] — Ratio (Cfed/C) of plasma 3TC has been presented

57. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP): Part 1 and 2
Description: SBP and DBP were measured in the supine or semi-supine position after 5 minutes rest. The Baseline value was considered to be the participant's last available assessment prior to time of the first dose. Change from Baseline was defined as post dose visit value minus Baseline value. Data for SBP and DBP for Part 1 and 2 is presented.
Time Frame: Up to Day 31 in Part 1 and Part 2
Population: Safety Population comprised of all participants who were enrolled in the study and received at least one dose of study drug. Only those participants available at the specified time points were analyzed represented by n=X,X,X,X,X,X in the category titles.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Groups:
- Part 1- A: DTG 50 mg + EPIVIR 300 mg: Participants received a single oral dose of DTG 50 mg and EPIVIR 300 mg tablet(s) at the same time with 240 mL of water in Periods 1 and 2 of Part 1. Treatments were administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
- Part 1- B: DTG 50 mg/ 3TC 300 mg Monolayer FDC: Participants received a single oral dose of DTG 50 mg and 3TC 300 mg monolayer FDC tablet formulation in Periods 1 and 2 of Part 1. Treatment was administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
- Part 1-Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed: Participants received DTG 50 mg and 3TC 300 mg monolayer FDC tablet formulation (Product Code AH). Treatment was administered with high fat meal. There was a washout period of at least 7 days (-4 hours) between each dose of the study drug.
- Part 2- A: DTG 50 mg + EPIVIR 300 mg: Participants received a single oral dose of DTG 50 mg and EPIVIR 300 mg tablet(s) at the same time with 240 mL of water in Periods 1 and 2 of Part 2. Treatments were administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
- Part 2-C: DTG 50 mg and 3TC 300 mg Bilayer FDC: Participants received a single oral dose of DTG 50 mg and 3TC 300 mg bilayer FDC tablet formulation in Periods 1 and 2 of Part 2. Treatment was administered in the fasted state after at least 10 hours of fasting. There was a washout period of at least 7 days between each dose of the study drug.
- Part 2-Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed: Participants received a single oral dose of DTG 50 mg and 3TC 300 mg bilayer FDC tablet formulation along with a high fat meal in Period 3 of Part 2.
Arm/Group | Part 1- A: DTG 50 mg + EPIVIR 300 mg | Part 1- B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Part 1-Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed | Part 2- A: DTG 50 mg + EPIVIR 300 mg | Part 2-C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Part 2-Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 75 | 76 | 16 | 75 | 75 | 16
Millimeters of mercury
  DBP,4 hour,n=75,76,16,75,75,16 | 0.1 (5.85) | 0.2 (5.24) | -2.1 (4.19) | -0.5 (4.09) | -0.3 (5.71) | 0.0 (4.86)
  DBP,Day 2,n=74,75,16,75,75,16: number analyzed (Participants) | 74 | 75 | 16 | 75 | 75 | 16
  DBP,Day 2,n=74,75,16,75,75,16 | -0.3 (5.53) | -0.9 (6.14) | 0.4 (5.32) | -1.7 (4.87) | -1.1 (4.99) | 3.1 (5.37)
  DBP,Day 3,n=74,75,16,75,75,16: number analyzed (Participants) | 74 | 75 | 16 | 75 | 75 | 16
  DBP,Day 3,n=74,75,16,75,75,16 | 3.2 (6.83) | 2.7 (5.95) | 1.3 (5.19) | 1.7 (5.74) | 1.2 (6.09) | 3.4 (5.76)
  DBP,Day 4,n=73,75,16,75,75,16: number analyzed (Participants) | 73 | 75 | 16 | 75 | 75 | 16
  DBP,Day 4,n=73,75,16,75,75,16 | 7.4 (6.47) | 5.4 (6.64) | 6.1 (4.22) | 4.9 (6.51) | 5.3 (6.11) | 8.3 (6.94)
  SBP,4 hour,n=75,76,16,75,75,16 | 1.5 (6.12) | 0.6 (5.94) | -0.8 (5.49) | 0.0 (5.04) | 0.5 (7.21) | 1.0 (7.28)
  SBP,Day 2,n=74,75,16,75,75,16: number analyzed (Participants) | 74 | 75 | 16 | 75 | 75 | 16
  SBP,Day 2,n=74,75,16,75,75,16 | -0.5 (6.88) | -1.4 (6.05) | 0.4 (3.91) | -1.5 (5.10) | -1.7 (7.12) | 1.9 (8.06)
  SBP,Day 3,n=74,75,16,75,75,16: number analyzed (Participants) | 74 | 75 | 16 | 75 | 75 | 16
  SBP,Day 3,n=74,75,16,75,75,16 | 4.0 (6.67) | 2.7 (6.15) | 2.9 (4.84) | 1.9 (7.28) | 1.6 (7.50) | 2.3 (7.73)
  SBP,Day 4,n=73,75,16,75,75,16: number analyzed (Participants) | 73 | 75 | 16 | 75 | 75 | 16
  SBP,Day 4,n=73,75,16,75,75,16 | 8.2 (8.09) | 7.5 (8.43) | 7.0 (5.80) | 7.0 (8.86) | 7.2 (8.72) | 7.6 (8.42)

58. Secondary Outcome: Change From Baseline in Heart Rate (HR): Part 1 and 2
Description: HR was measured in the supine or semi-supine position after 5 minutes rest. The Baseline value was considered to be the participant's last available assessment prior to time of the first dose. Change from Baseline was defined as post dose visit value minus Baseline value. Data for HR for Part 1 and 2 is presented.
Time Frame: Up to Day 31 in Part 1 and Part 2
Population: Safety Population. Only those participants available at the specified time points were analyzed represented by n=X,X,X,X,X,X in the category titles.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1- A: DTG 50 mg + EPIVIR 300 mg | Part 1- B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Part 1-Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed | Part 2- A: DTG 50 mg + EPIVIR 300 mg | Part 2-C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Part 2-Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 75 | 76 | 16 | 75 | 75 | 16
Beats per minute
  4 hour,n=75,76,16,75,75,16 | 0.6 (5.49) | 0.4 (4.25) | 4.9 (3.84) | 0.1 (5.25) | -0.3 (5.43) | 3.0 (3.22)
  Day 2,n=74,75,16,75,75,16: number analyzed (Participants) | 74 | 75 | 16 | 75 | 75 | 16
  Day 2,n=74,75,16,75,75,16 | 2.2 (5.53) | 1.9 (4.60) | 2.9 (4.17) | 1.6 (5.48) | 0.6 (5.74) | 1.6 (5.44)
  Day 3,n=74,75,16,75,75,16: number analyzed (Participants) | 74 | 75 | 16 | 75 | 75 | 16
  Day 3,n=74,75,16,75,75,16 | 5.1 (8.15) | 6.0 (6.35) | 5.8 (6.80) | 5.3 (7.23) | 3.8 (7.13) | 7.7 (10.42)
  Day 4,n=73,75,16,75,75,16: number analyzed (Participants) | 73 | 75 | 16 | 75 | 75 | 16
  Day 4,n=73,75,16,75,75,16 | 7.5 (9.28) | 8.9 (7.68) | 9.6 (9.15) | 8.9 (8.31) | 6.1 (8.39) | 9.5 (10.10)

59. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs): Part 1 and 2
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinaemia were categorized as SAE. Participants having any AE or SAE are presented.
Time Frame: Up to Week 11
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- A: DTG 50 mg + EPIVIR 300 mg | Part 1- B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Part 1-Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed | Part 2- A: DTG 50 mg + EPIVIR 300 mg | Part 2-C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Part 2-Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
Number analyzed (Participants) | 75 | 76 | 16 | 75 | 75 | 16
Participants
  AEs | 14 | 18 | 1 | 15 | 12 | 1
  SAEs | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the start of study treatment until the follow-up contact (Up to 11 weeks)
Description: Safety Population comprised of all participants who were enrolled in the study and received at least one dose of study drug.
Arm/Group | Part 1- A: DTG 50 mg + EPIVIR 300 mg | Part 1- B: DTG 50 mg/ 3TC 300 mg Monolayer FDC | Part 1-Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed | Part 2- A: DTG 50 mg + EPIVIR 300 mg | Part 2-C: DTG 50 mg and 3TC 300 mg Bilayer FDC | Part 2-Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76 | 0/16 | 0/75 | 0/75 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/76 | 0/16 | 0/75 | 0/75 | 0/16
Other Adverse Events (participants affected / at risk) | 2/75 | 5/76 | 1/16 | 8/75 | 6/75 | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1- A: DTG 50 mg + EPIVIR 300 mg (N=75) | Part 1- B: DTG 50 mg/ 3TC 300 mg Monolayer FDC (N=76) | Part 1-Bfed: DTG 50 mg and 3TC 300 mg Monolayer FDC Fed (N=16) | Part 2- A: DTG 50 mg + EPIVIR 300 mg (N=75) | Part 2-C: DTG 50 mg and 3TC 300 mg Bilayer FDC (N=75) | Part 2-Cfed: DTG 50 mg and 3TC 300 mg Bilayer FDC Fed (N=16)
Headache (Nervous system disorders) | 2 | 5 | 1 | 8 | 6 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT03078556/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT03078556/SAP_001.pdf